CLINICAL TRIAL: NCT01255072
Title: Repetitive Transcranial Magnetic Stimulation in Elderly Depressed: Neuronavegated Study
Brief Title: rTMS in Elderly Depressed:Neuronavegated Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Bianca Boura Bellini, Department and Institute of Psychiatry, General Hospital, University of São Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBellini - 0996/07
Record Dates: First submitted 2010-12-03; First posted 2010-12-07 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2007-05

CONDITIONS: DEPRESSION
Keywords: TMS; elderly; depression; neuronavegation; neurocognition
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS + placebo (Active Comparator): Patients, free from medication for at least one week (washout of 3 weeks for fluoxetine users) will receive 20 sessions of active rTMS delivered to the left Dorsolateral PreFrontal Cortex. Each patient will take placebo pills for 60 day,starting parallel on the first rTMS day.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation
- SHAM (Sham Comparator): Patients, free from medication at least for one week (washout of 3 weeks for fluoxetine users)receiving 20 sessions of Sham TMS delivered to the left dordolateral prefrontal cortex, at the same time this washed out of antidepressives patients start taking Citalopram 20mg/day, for 60 days.
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — 20 Sham daily sessions:25 trains, 10seconds at 5Hz, train interval of 25 seconds (time off). Target: left dorsolateral prefrontal cortex.
  Other Names: Sham TMS
  Arms: SHAM
Procedure: Repetitive Transcranial Magnetic Stimulation — 20 daily sessions: each one with 25 trains of 10seconds at 5Hz, train interval of 25 seconds (time off), pulse intensity corrected based on atrophy degree by a specific correction formule. Target: left dorsolateral prefrontal cortex.
  Other Names: TMS
  Arms: Active rTMS + placebo

SUMMARY:
This double-blind, controlled and randomized study intents to investigate the antidepressive response of rTMS on the elderly population.This is the first neuronavegated pulse intensity corrected study of rTMS in elderly depressed patients.

DETAILED DESCRIPTION:
Most part of the studies uses samples of severe depressive patients with refractoriness and/or psychotic symptoms, which leave lacuna about the effects on depressive disorder with low or moderate scores. The literature is poor about the use of Repetitive Transcranial Magnetic Stimulation (rTMS) in the old age population.Therefore, we chose this group to research for the antidepressive effect of TMS; other interests are to identify modifications in the magnetic resonance imaging, evaluate cognitive functions and to verify the occurrence of collateral effects and safety use for this specific population.

ELIGIBILITY:
METHODS:Forty patients with the following criteria:

Inclusion Criteria

* Patients who meet criteria for Major Depressive Episode (MDE) (DSM-IV, 1994; SCID-P, 1994);
* Severity of the episode of mild to moderate
* Aged between 60 and 75 years;
* Both genders;
* In case of previous depressive episode, complete remission of the same for at least 6 weeks as measured by the clinical history;
* washed out of psychotropic drugs for one week, including antidepressants; except fluoxetine, which must have three week interval;
* Granting a written informed consent to participate in the study (Annex II)

Exclusion Criteria:

* metallic cerebral implants
* history of severe trauma or brain injury
* organic brain disease
* severe somatic disease
* history of other psychiatric diseases
* history of Epilepsy
* Non cooperating patients

Scales and Tests of clinical evaluation:

1. Hamilton Depression Rating Scale-17 items
2. Geriatric Depression Scale (GDS)
3. Mini Mental State Examination
4. Clock Drawing Test
5. Clinical Dementia Rating
6. Visual Analogue Scale
7. Clinical Global Impression.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of the depressive symptomatology on 50% in relation to the initial scored by HAM-D/17 scale, or complete remission of the episode, defined as HAM-D/17 score ≤ 7 at the end of the treatment. | 30 months
  evaluation also by Geriatric Depression Scale (GDS)

SECONDARY OUTCOMES:
Reduction of the depressive symptomatology on 50% in relation to the initial scored by HAM-D/17 scale, or complete remission of the episode, defined as HAM-D/17 score ≤ 7 at the end of the treatment. | 30 months
  recruting

CONTACTS AND LOCATIONS:
Overall Officials: Bianca B. Bellini, Principal Investigator — Department and Institute os Psychiatry, General Hospital, University Of São Paulo
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of Sao Paulo medical school, São Paulo, São Paulo, Brazil